CLINICAL TRIAL: NCT00002953
Title: A Radomized Trial of Epirubicin & Cyclophosphamide vs. Epirubicin & Paclitaxel in the Treatment of Women With Metastatic Breast Cancer
Brief Title: Epirubicin and Cyclophosphamide Compared With Epirubicin and Paclitaxel in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065426; MRC-UKCCCR-AB01; EU-97002
Record Dates: First submitted 1999-11-01; First posted 2004-07-07 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2005-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Epirubicin; Paclitaxel

INTERVENTIONS:
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of epirubicin and cyclophosphamide with epirubicin and paclitaxel in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the activity and toxicity of epirubicin and cyclophosphamide with that of epirubicin and paclitaxel in patients with metastatic breast cancer.

OUTLINE: Patients are randomized to receive either epirubicin and cyclophosphamide or epirubicin and paclitaxel. Each drug combination is given every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 704 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven carcinoma of the breast with metastases No CNS metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Not specified Menopausal status: Not specified Sex: Female Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.25 times upper limit of normal (ULN) SGOT and SGPT no greater than 2 times ULN (no greater than 5 times ULN with liver metastases) Renal: Not specified Cardiovascular: Ejection fraction within normal range No history of cardiac disease including myocardial infarction, cardiac failure and angina Other: Not pregnant No prior or concurrent malignancy that is likely to interfere with protocol treatments or comparisons

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy other than adjuvant No prior high dose adjuvant chemotherapy requiring transplantation Cumulative dose of doxorubicin no greater than 300 mg/m2 permitted Cumulative dose of epirubicin no greater than 400 mg/m2 permitted At least 6 months since prior anthracyclines Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 704 (Estimated)
Dates: Start 1996-12; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Carmichael, MD, PhD, Study Chair — Nottingham City Hospital
Locations (19):
- Groote Schuur Hospital, Cape Town, Cape Town, South Africa
- United Kingdom (18):
  - University Birmingham, Birmingham, England
  - Bristol Royal Hospital for Sick Children, Bristol, England
  - Bristol Oncology Centre, Bristol, England
  - Derbyshire Royal Infirmary, Derby, England
  - Cookridge Hospital, Leeds, England
  - University Hospitals of Leicester, Leicester, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Hospital, Northwood, England
  - Norfolk & Norwich Hospital, Norwich, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Royal Marsden Hospital, Sutton, England
  - Southend General Hospital, Westcliff-on-Sea, England
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - Royal Preston Hospital, Preston

REFERENCES:
- [Result] Langley RE, Carmichael J, Jones AL, Cameron DA, Qian W, Uscinska B, Howell A, Parmar M. Phase III trial of epirubicin plus paclitaxel compared with epirubicin plus cyclophosphamide as first-line chemotherapy for metastatic breast cancer: United Kingdom National Cancer Research Institute trial AB01. J Clin Oncol. 2005 Nov 20;23(33):8322-30. doi: 10.1200/JCO.2005.01.1817. PMID 16293863
- [Result] Carmichael J: UKCCCR trial of epirubicin and cyclophosphamide (EC) vs. epirubicin and taxol (ET) in the first line treatment of women with metastatic breast cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-84, 2001.
- [Result] Carmichael J: UKCCCR trial of epirubucin and cyclophosphamide (EC) versus epirubicin and taxol (ET) in the first line treatment of women with metastatic breast cancer (MBC). [Abstract] Br J Cancer 85 (suppl 1): A-CT6, 2, 2001.